CLINICAL TRIAL: NCT02622178
Title: Sensitivity and Specificity of the NOVA-DN VEP Protocol and a Novel Analysis of Optical Coherence Tomography Images for Glaucoma Diagnosis
Brief Title: How Accurately Does the Diopsys Visual Evoked Potential (VEP) Vision Testing System Detect Glaucoma?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-125E
Record Dates: First submitted 2015-08-06; First posted 2015-12-04 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Glaucoma Diagnosis
MeSH Terms: interventions — Tomography, Optical Coherence; Evoked Potentials, Visual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Healthy Subjects (Experimental): 42 Healthy subjects with intraocular pressure less than 22 millimeters of mercury (mmHg), normal appearing optic discs and retinal nerve fiber layer, normal optical coherence technology (RNFL thickness) and normal visual field results in both eyes. Participants will have optical coherence tomography (OCT) and Diopsys visual evoked potential testing (VEP).
  Interventions: Diagnostic Test: Optical Coherence Tomography; Diagnostic Test: Visual evoked potential
- Glaucoma Suspects (Experimental): 45 Glaucoma suspects with glaucomatous appearance optic discs and/or thin retinal nerve fiber layer in at least one eye, normal optical coherence technology (RNFL thickness) and normal visual field results in both eyes. Participants will have optical coherence tomography (OCT) and Diopsys visual evoked potential testing (VEP).
  Interventions: Diagnostic Test: Optical Coherence Tomography; Diagnostic Test: Visual evoked potential
- Glaucoma Patients (Experimental): 49 Glaucoma patients with repeatable abnormal visual fields, glaucomatous optic disc appearance (those with cup to disc ratio greater than 0.7, rim thinning or Retinal Nerve Fiber Layer defects indicative of glaucoma) and/or repeatable intra-ocular pressure of 23 mmHg or higher, in at least one eye. Participants will have optical coherence tomography (OCT) and Diopsys visual evoked potential testing (VEP).
  Interventions: Diagnostic Test: Optical Coherence Tomography; Diagnostic Test: Visual evoked potential

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — Optical coherence tomography (OCT) is a noninvasive imaging modality that provides micrometer-scale resolution.It has been revolutionized in recent years by exploitation of Fourier domain (FD) techniques, which have a significant sensitivity advantage over traditional time domain (TD) OCT. In spectral-domain (SD-OCT) the reference mirror is stationary, and OCT signal is acquired using a spectrometer as detector or by varying the wavelength of the light source.
  Other Names: OCT
Diagnostic Test: Visual evoked potential — Visual evoked potential is a means of objectively testing visual field by viewing a computer monitor at 1 meter with a square black/white checkerboard pattern reversal stimulus. Electrodes are placed on the head and face to monitor Electroencephalogram (EEG) activity during testing. Output parameters from VEP system include amplitude and latency measures for each stimuli.
  Other Names: VEP

SUMMARY:
Evaluate sensitivity and specificity of NOVA-DN visually evoked potentials (VEP) protocol and new software method (Corda) for glaucoma detection using optical coherence tomography (OCT) images to differentiate between normal subjects and glaucoma suspects.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the ability of NOVA-DN VEP protocol and Corda parameters to discriminate between healthy eyes and eyes with early to moderate glaucomatous visual field loss. We will evaluate measurements of the NOVA-DN VEP protocol, Corda software and Cirrus spectral domain (SD) OCT software in order to compare and correlate.

Hypotheses is that NOVA-DN VEP protocol and Corda analysis results in a high sensitivity, specificity and area under the Receiver Operating Characteristic (ROC) curves (ROC area) for glaucoma detection. Second hypothesis is NOVA-DN VEP protocol and Corda parameters can differentiate between normal and glaucoma suspects.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Healthy Subjects

* intraocular pressure less than 22 millimeters of mercury (mmHg)
* normal appearing optic discs and retinal nerve fiber layer (RNFL)
* normal optical coherence tomography (OCT) RNFL thickness
* normal visual field (VF) results in both eyes.

Group 2: Glaucoma Suspects

* glaucomatous appearance of optic discs and/or RNFL in at least one eye
* normal OCT
* normal VF results in both eyes.

Group3: Glaucoma Patients

* Glaucomatous optic disc appearance (cup to disc ratio, rim thinning or RNFL defects)
* Repeatable intraocular pressure (IOP) of 23 mmHg or more, in at least one eye
* Repeatable abnormal VF tests

Exclusion Criteria:

* inability to perform reliable VF or OCT
* visual acuity worse than 20/40
* refractive error greater than +/-5.00 diopters sphere, greater than +/- 3.00 diopers cylinder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L J Katz, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Manuscript has been published.

REFERENCES:
- [Result] Waisbourd M, Gensure RH, Aminlari A, Shah SB, Khanna N, Sood N, Molineaux J, Gonzalez A, Myers JS, Katz LJ. Short-duration transient visual evoked potentials and color reflectivity discretization analysis in glaucoma patients and suspects. Int J Ophthalmol. 2017 Feb 18;10(2):254-261. doi: 10.18240/ijo.2017.02.12. eCollection 2017. PMID 28251085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Glaucoma patients, suspects and healthy subjects were recruited between 2011 and 2012 in the Glaucoma Service at Wills Eye Hospital, Philadelphia, Pennsylvania, USA.
Groups:
- Healthy Subjects: 42 Healthy subjects with intraocular pressure less than 22 millimeters of mercury (mmHg), normal optic discs and retinal nerve fiber layer, normal optical coherence technology (RNFL thickness) and normal visual fields in both eyes will have optical coherence tomography (OCT) imaging and visual evoked potential (VEP) testing.
  Optical coherence tomography (OCT), noninvasive imaging, provides micrometer-scale resolution. It utilizes Fourier domain (FD) techniques, with sensitivity advantage over traditional time domain (TD).
  Visual evoked potential (VEP) objectively tests visual field by viewing a monitor at 1 meter of square black/white checks with electrodes on back of head where vision is processed.
- Glaucoma Suspects: 45 Glaucoma suspects with glaucomatous optic discs and/or thin retinal nerve fiber layer in at least one eye, normal optical coherence technology and normal visual field results will have optical coherence tomography (OCT) imaging and visual evoked potential (VEP) testing.
  Optical coherence tomography (OCT), noninvasive imaging, provides micrometer-scale resolution. It utilizes Fourier domain (FD) techniques, with sensitivity advantage over traditional time domain (TD).
  Visual evoked potential (VEP) objectively tests visual field by viewing a monitor at 1 meter of square black/white checks with electrodes on back of head where vision is processed.
- Glaucoma Patients: 49 Glaucoma patients with repeatable abnormal visual fields, glaucomatous optic disc (those with cup to disc ratio greater than 0.7, rim thinning or Retinal Nerve Fiber Layer defects indicative of glaucoma) and/or repeatable intra-ocular pressure of 23 mmHg or higher, in at least one eye will have optical coherence tomography (OCT) imaging and visual evoked potential (VEP) testing.
  Optical coherence tomography (OCT), noninvasive imaging, provides micrometer-scale resolution. It utilizes Fourier domain (FD) techniques, with sensitivity advantage over traditional time domain (TD).
  Visual evoked potential (VEP) objectively tests visual field by viewing a monitor at 1 meter of square black/white checks with electrodes on back of head where vision is processed.
Period: Overall Study
Arm/Group | Healthy Subjects | Glaucoma Suspects | Glaucoma Patients
Started | 42 | 45 | 49
Completed | 42 | 45 | 49
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Subjects: 42 Healthy subjects with intraocular pressure less than 22 millimeters of mercury (mmHg), normal optic discs and retinal nerve fiber layer, normal optical coherence technology (RNFL thickness) and normal visual fields in both eyes for optical coherence tomography (OCT) and visual evoked potential testing (VEP).
  Optical Coherence Tomography: Optical coherence tomography (OCT) is a noninvasive imaging modality that provides micrometer-scale resolution.It has been revolutionized in recent years by exploitation of Fourier domain (FD) techniques, which have a significant sensitivity advantage over traditional time domain (TD) OCT. In spectral-domain (SD-OCT) the reference mirror is stationary, and OCT signal is acquired using a spectrometer as detector or by varying the wavelength of the light source.
  Visual evoked potential: Visual evoked potential is a means of objectively testing visual field by viewing a computer monitor at 1 meter wit
- Glaucoma Suspects: 45 Glaucoma suspects with glaucomatous optic discs and/or thin retinal nerve fiber layer in at least one eye, normal optical coherence technology and normal visual field results will have optical coherence tomography and visual evoked potential.
  Optical Coherence Tomography: Optical coherence tomography (OCT) is a noninvasive imaging modality that provides micrometer-scale resolution.It has been revolutionized in recent years by exploitation of Fourier domain (FD) techniques, which have a significant sensitivity advantage over traditional time domain (TD) OCT. In spectral-domain (SD-OCT) the reference mirror is stationary, and OCT signal is acquired using a spectrometer as detector or by varying the wavelength of the light source.
  Visual evoked potential: Visual evoked potential is a means of objectively testing visual field by viewing a computer monitor at 1 meter with a square black/white check
- Glaucoma Patients: 49 Glaucoma patients with repeatable abnormal visual fields, glaucomatous optic disc (those with cup to disc ratio greater than 0.7, rim thinning or Retinal Nerve Fiber Layer defects indicative of glaucoma) and/or repeatable intra-ocular pressure of 23 mmHg or higher, in at least one eye will have optical coherence tomography and visual evoked potential.
  Optical Coherence Tomography: Optical coherence tomography (OCT) is a noninvasive imaging modality that provides micrometer-scale resolution.It has been revolutionized in recent years by exploitation of Fourier domain (FD) techniques, which have a significant sensitivity advantage over traditional time domain (TD) OCT. In spectral-domain (SD-OCT) the reference mirror is stationary, and OCT signal is acquired using a spectrometer as detector or by varying the wavelength of the light source.
  Visual evoked potential: Visual evoked potential is a means of objectively testing visu
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects | Glaucoma Suspects | Glaucoma Patients | Total
Number analyzed (Participants) | 42 | 45 | 49 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 33 | 95
  >=65 years | 12 | 13 | 16 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 27 | 57
  Male | 30 | 27 | 22 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 24 | 21 | 56
  White | 30 | 13 | 27 | 70
  More than one race | 0 | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 45 | 49 | 136

OUTCOME MEASURES:

1. Primary Outcome: Visual Evoked Potential (VEP)
Description: Diopsys Visual evoked potential (VEP) (Diopsys, Inc. Pine Brook, NJ) is used to objectively measure the functional responses of the entire visual pathway from the anterior segment of the eye to the visual cortex. This is the strength of the signal recorded from the back of the head near where vision is processed in the brain while a visual stimulus is presented to patient.
Time Frame: 1 examination, one hour
Population: measurement is amplitude in microvolts (uV), the peak strength of the signal, when presented with low contrast stimuli
Measure: Mean (Standard Deviation); unit: microvolts (uV) (amplitude)
Groups:
- Glaucoma Patients: 49 Glaucoma patients with repeatable abnormal visual fields, glaucomatous optic disc (cup to disc ratio greater than 0.7, rim thinning or glaucomatous Retinal Nerve Fiber Layer defects) and/or repeatable intra-ocular pressure of 23 mmHg or higher, in at least one eye will have optical coherence tomography (OCT) imaging and visual evoked potential (VEP) testing.
  Optical coherence tomography (OCT), noninvasive imaging, provides micrometer-scale resolution. It utilizes Fourier domain (FD) techniques, with sensitivity advantage over traditional time domain (TD).
  Visual evoked potential (VEP) objectively tests visual field by viewing a monitor at 1 meter of square black/white checks with electrodes on back of head where vision is processed.
Arm/Group | Healthy Subjects | Glaucoma Suspects | Glaucoma Patients
Number analyzed (Participants) | 42 | 45 | 49
microvolts (uV) (amplitude) | 6.7 (3.3) | 7.1 (3.9) | 4.1 (2.7)

2. Secondary Outcome: Retinal Nerve Fiber Layer Thickness
Description: Optical coherence tomography (OCT) images provide measurement of the retinal nerve fiber layer thickness in microns.
Time Frame: 1 examination, one hour
Measure: Mean (Standard Deviation); unit: microns (thickness)
Arm/Group | Healthy Subjects | Glaucoma Suspects | Glaucoma Patients
Number analyzed (Participants) | 42 | 45 | 49
microns (thickness) | 95.1 (8.7) | 87.5 (13.4) | 71.2 (12.1)

ADVERSE EVENTS:
Time Frame: 1 examination, one hour
Description: No adverse or serious adverse events were reported during this 1 examination, one hour study.
Arm/Group | Healthy Subjects | Glaucoma Suspects | Glaucoma Patients
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/45 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45 | 0/49
Other Adverse Events (participants affected / at risk) | 0/42 | 0/45 | 0/49

LIMITATIONS AND CAVEATS:
Small sample size. Participants were all recruited from one large urban setting. Age difference between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No